CLINICAL TRIAL: NCT00296634
Title: A Phase I-II, Randomized, Controlled, Dose-Ranging Study of the Safety, Reactogenicity, and Immunogenicity of Intramuscular Inactivated Influenza A/H5N1 Vaccine Given Alone or With Aluminum Hydroxide to Healthy Adults
Brief Title: H5 Vaccine Alone or With Adjuvant in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Robert Johnson, HHS/NIAID/DMID
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 05-0127
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2008-09

CONDITIONS: Influenza
Keywords: H5N1, Influenza, vaccine
MeSH Terms: conditions — Influenza, Human; Influenza in Birds | interventions — Aluminum Hydroxide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental): 45 microgram dose Hemagglutinin (HA), 120 subjects receiving Aluminum hydroxide and 120 not receiving Aluminum hydroxide.
  Interventions: Drug: Aluminum hydroxide; Biological: Inactivated Influenza A/H5N1 Vaccine (sanofi pasteur pre-adsorbed)
- 2 (Experimental): 15 microgram dose HA, 60 subjects receiving Aluminum hydroxide and 60 not receiving Aluminum hydroxide.
  Interventions: Drug: Aluminum hydroxide; Biological: Inactivated Influenza A/H5N1 Vaccine (sanofi pasteur pre-adsorbed)
- 4 (Experimental): 3.75 microgram dose HA, 60 subjects receiving Aluminum hydroxide and 60 not receiving Aluminum hydroxide.
  Interventions: Drug: Aluminum hydroxide; Biological: Inactivated Influenza A/H5N1 Vaccine (sanofi pasteur pre-adsorbed)
- 3 (Experimental): 7.5 microgram dose HA, 60 subjects receiving Aluminum hydroxide and 60 not receiving Aluminum hydroxide.
  Interventions: Drug: Aluminum hydroxide; Biological: Inactivated Influenza A/H5N1 Vaccine (sanofi pasteur pre-adsorbed)

INTERVENTIONS:
Drug: Aluminum hydroxide — Aluminum hydroxide adjuvant at 1200 mcg/mL.
Biological: Inactivated Influenza A/H5N1 Vaccine (sanofi pasteur pre-adsorbed) — Inactivated monovalent subvirion influenza H5N1 vaccine produced with and without Aluminum hydroxide adjuvant. All formulations of the H5N1 vaccine are supplied in a unit dose (0.5 mL) vial as a sterile solution for intramuscular injection. Vaccine with adjuvant is a turbid liquid whitish-grey in color. Vaccine without adjuvant is essentially clear and slightly opalescent in color.

SUMMARY:
This randomized, controlled, double-blinded, dose-ranging, Phase I-II study in 600 healthy adults, 18 to 49 years old, is designed to investigate the safety, reactogenicity, and dose-related immunogenicity of an investigational inactivated influenza A/H5N1 virus vaccine when given alone or combined with aluminum hydroxide. A secondary goal is to guide selection of vaccine dosage levels for expanded Phase II trials based on reactogenicity and immunogenicity profiles. This dose optimization will be applied to both younger and older subject populations in subsequent studies. Subjects who meet the entry criteria for the study will be enrolled at one of 4 study sites and will be randomized into one of 8 groups to receive 2 doses of influenza A/H5N1 vaccine containing 3.75, 7.5, 15, or 45 mcg of HA with or without aluminum hydroxide adjuvant by intramuscular injection. Participants may be involved in study related procedures for up to 8 months.

DETAILED DESCRIPTION:
This randomized, controlled, double-blinded, dose-ranging, Phase I/II study in healthy adults, 18 to 49 years old, is designed to investigate the safety, reactogenicity, and dose-related immunogenicity of an investigational inactivated influenza A/H5N1 virus vaccine when given alone or combined with aluminum hydroxide. The primary objectives are to: determine the dose-related safety of subvirion-inactivated H5N1 vaccine adjuvanted with aluminum hydroxide in healthy adults; determine the potential for aluminum hydroxide to enhance the immune response to subvirion-inactivated H5N1 vaccine in healthy adults approximately 1 month following receipt of 2 doses of vaccine; and provide information for the selection of the best dosage level for further studies. The secondary objective is to evaluate dose-related immunogenicity and the percent of subjects responding approximately 1 and 7 months after the first vaccination. This dose optimization will be applied to both younger and older subject populations in subsequent studies. Subjects who meet the entry criteria for the study will be randomized into 8 groups to receive 2 doses of influenza A/H5N1 vaccine containing 3.75, 7.5, 15, or 45 mcg of hemagglutinin (HA) with or without aluminum hydroxide adjuvant by intramuscular (IM) injection (N=60 or 120/vaccine dose group). The first vaccination will occur on Day 0. Symptoms and signs will be assessed in the clinic for at least 15 minutes after inoculation, and the subjects will maintain a memory aid to record oral temperature and systemic and local adverse events (AEs) for 7 days after each immunization. Subjects will be encouraged to take their temperature around the same time each day. All subjects will return to the clinic 2 days and 8 days after each vaccination for assessment of adverse events (AEs) and concomitant medications and targeted physical examination (if indicated). Memory aids will be reviewed at each visit. Approximately Day 28 after the first vaccination, subjects will return to the clinic for blood sample collection and safety follow-up, followed by a second vaccination. Approximately 56 days after first immunization (or about 28 days after the second vaccination), subjects will return to the clinic for immunogenicity blood sample collection, AE and concomitant medication assessment, and targeted physical examination (if indicated). At approximately Day 208 (7 months after the first vaccination), subjects will return to the clinic for a final immunogenicity blood sample collection and for follow-up (which includes a targeted physical examination [if indicated]). Blood samples collected prior to each vaccination and on Days 56 and 208 after the first vaccination will be tested in a central laboratory for the levels of neutralizing and HAI antibodies. The primary outcome measures will be the frequencies and severities of AEs in each group and the proportions of subjects who achieve a serum neutralizing antibody titer of greater than or equal to 1:40 against the influenza A/H5N1 virus on Day 56. Serum HAI and neutralizing antibody responses (including frequencies of 4 fold or greater rise in titers; geometric mean titers; and proportions of subjects achieving putative protective titers of neutralizing antibody 1 month after each dose of vaccine and 7 months after first dose) also will be assessed. Although the correlate of protection for infections caused by influenza A/H5N1 viruses in humans is unknown, a serum neutralizing antibody titer of greater than or equal to 1:40 may be considered protective, based on limited data regarding the levels of serum neutralizing antibody present in serum samples collected from humans who survived infections caused by influenza A/H5N1 viruses. This study is linked to DMID protocol 07-0022.

ELIGIBILITY:
Inclusion Criteria:

* Are males or nonpregnant females between the ages of 18 and 49 years, inclusive.
* Agree to practice adequate contraception (i.e., barrier methods, abstinence, intrauterine devices, and licensed hormonal methods) for the entire study period if they are females of childbearing potential (not surgically sterile or postmenopausal for greater than or equal to 1 year).
* Are in good health as determined by vital signs, medical history to ensure stable medical condition, and targeted physical examination based on medical history.
* Are able to understand and comply with planned study procedures.
* Provide written informed consent prior to initiation of any study procedures.

Stable medical condition - no change in prescription medication, dose, or frequency of medication in the last 3 months and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months. Any change that is due to change of health care provider, insurance company etc, or that is done for financial reasons, as long as in the same class of medication will not be considered a violation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome will not be considered a violation of this inclusion criterion.

Exclusion Criteria:

* Have a known allergy to eggs or other components of the vaccine (including gelatin, formaldehyde, octoxinol, thimerosal, aluminum hydroxide, and chicken protein).
* Have a positive urine or serum pregnancy test prior to vaccination (if female of childbearing potential) or are women who are breastfeeding.
* Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months.
* Have an active neoplastic disease or a history of any hematologic malignancy.
* Have long-term use of oral steroids, parenteral steroids, or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (Nasal and topical steroids are allowed.).
* Have a diagnosis of schizophrenia, Bi-polar disease or other major psychiatric diagnosis.
* Have been hospitalized for psychiatric illness, history of suicide attempt or confinement for danger to self or others.
* Are receiving psychiatric drugs (aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, chlorprothixene, chlorpromazine, perphenazine, trifluopromazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate). Subjects who are receiving a single antidepressant drug and stable for at least 3 months prior to enrollment, without de-compensating symptoms will be allowed to be enrolled in the study.
* Have a history of receiving immunoglobulin or other blood product within the 3 months prior to vaccination in this study.
* Have received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to vaccination in this study.
* Have an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses (This includes, but is not limited to, known chronic liver disease, significant renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients.).
* Have a history of severe reactions following immunization with contemporary influenza virus vaccines.
* Have an acute illness, including an oral temperature greater than 100.4 degrees F, within 1 week of vaccination.
* Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to vaccination in this study or expect to receive an experimental agent during the 7-month study period.
* Have any condition that would, in the opinion of the site investigator, place them at an unacceptable risk of injury or render them unable to meet the requirements of the protocol.
* Participated in an influenza A/H5 vaccine study in the past in a group receiving vaccine (but does not exclude documented placebo recipients).
* Have a known active human immunodeficiency virus, hepatitis B, or hepatitis C infection.
* Have a history of alcohol or drug abuse in the last 5 years.
* Planned to travel outside of the USA in the time between the first vaccination and 56 days following the first vaccination.
* Have a history of Guillain Barre syndrome.
* Have any condition that the investigator believes may interfere with successful completion of the study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2006-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Adverse event (AE) or serious adverse event (SAE) information (solicited in the clinic and via memory aids, concomitant medications, and periodic targeted physical assessments). | Adverse events will be collected through 28 days following the second dose of vaccine (approximately Day 56). Serious adverse events will be collected throughout the study through Day 208.
Proportion of subjects in each group achieving a serum neutralizing antibody titer of greater than or equal to 1:40 against the influenza A/H5N1 virus. | 28 days following second dose of vaccine.
Proportion of subjects in each dose group achieving a serum Hemagglutination Inhibition (HAI) antibody titer of greater than or equal to 1:40 against the influenza A/H5N1 virus. | 28 days following second dose of vaccine.
Geometric mean titer (GMT) and frequency of 4-fold or greater increases in neutralizing antibody titers in each group. | 28 days following second dose of vaccine.
Geometric mean titer (GMT) and frequency of 4-fold or greater increases in serum HAI antibody titers in each group. | 28 days after receipt of the second dose of vaccine.

SECONDARY OUTCOMES:
1 month after receipt of each dose, and 7 months after receipt of the first dose of vaccine. | 1 month after receipt of each dose, and 7 months after receipt of the first dose of vaccine.
Geometric mean titer (GMT) and the frequency of 4-fold or greater increases in serum HAI antibody titers. | 1 month after receipt of each dose, and 7 months after receipt of the first dose of vaccine.
Development of serum antibody responses against antigenically drifted variants of H5N1 influenza virus. | Blood samples for serum assays will be collected at day 0 and at days 28, 56, and 208 after the first immunization.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Maryland Baltimore, Baltimore, Maryland
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Derived] Keitel WA, Campbell JD, Treanor JJ, Walter EB, Patel SM, He F, Noah DL, Hill H. Safety and immunogenicity of an inactivated influenza A/H5N1 vaccine given with or without aluminum hydroxide to healthy adults: results of a phase I-II randomized clinical trial. J Infect Dis. 2008 Nov 1;198(9):1309-16. doi: 10.1086/592172. PMID 18808338